CLINICAL TRIAL: NCT02612987
Title: Internet-delivered Cognitive Behaviour Therapy for Adolescents With Co-morbid Insomnia Attending Children and Youth Psychiatry: An Open Trial
Brief Title: iCBT for Adolescents With Co-morbid Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Collaborators: Karolinska Institutet (Other); Uppsala University (Other)
Responsible Party: Principal Investigator, Vendela Zetterqvist, Ph D, licensed psychologist, Uppsala University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015/326
Record Dates: First submitted 2015-11-15; First posted 2015-11-24 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Dyssomnias
Keywords: CBT; Internet based
MeSH Terms: conditions — Dyssomnias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- iCBT (Experimental)
  Interventions: Behavioral: Internet-based Cognitive Behaviour Therapy (iCBT)

INTERVENTIONS:
Behavioral: Internet-based Cognitive Behaviour Therapy (iCBT)

SUMMARY:
Insomnia is a commonly reported comorbidity for adolescents with psychiatric conditions. It is well-known that insomnia can exacerbate the concurrent psychiatric symptom load. Treatment of insomnia has been extensively examined in adults, but studies with adolescents are sparse. The purpose of this pilot study is to assess the feasibility and efficacy of internet-based cognitive behavioral therapy for insomnia (iCBT) in outpatients of Children and Youth Psychiatry. Twenty-one adolescents will be recruited and receive 7 weeks of iCBT. Outcome will be measured at pre treatment, at post treatment and at a three months follow-up. Weekly assessments will also be made during treatment on primary outcome and a presumed process variable constructed for the purpose of this trial.

ELIGIBILITY:
Inclusion Criteria:

* To fulfill the diagnostic criteria for insomnia
* To have access to a computer with Internet connection
* No previous or ongoing CBT for insomnia
* No psychotropic medication or being on a stable dosage for at least six weeks before enrollment

Exclusion Criteria:

* Ongoing manic or psychotic episode
* Being at high risk of triggering manic or psychotic episode
* Ongoing sleep apnea

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2015-10; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI; Morin, 1993) | Pre treatment, weekly during treatment (e.g. from date of treatment start for seven weeks until treatment is terminated), post treatment (e.g. seven weeks after the patient has started treatment), 3 month follow-up
  Given that this is an intervention study we are assessing changes in outcome over time.

SECONDARY OUTCOMES:
The Core Consensus Sleep Diary (Core CSD; Carney et al., 2012) | Pre treatment, weekly during treatment (e.g. from date of treatment start for seven weeks until treatment is terminated), post treatment (e.g. seven weeks after the patient has started treatment), 3 month follow-up
  Given that this is an intervention study we are assessing changes in outcome over time.
Symptoms Checklist (SCL-90; Derogatis et al., 1994) | Pre treatment, post treatment (e.g. seven weeks after the patient has started treatment), 3 month follow-up
  Given that this is an intervention study we are assessing changes in outcome over time.
Montgomery-Åsberg Depression Rating Scale - Self report (MADRS-S; Svanborg & Åsberg, 1994) | Pre treatment, post treatment (e.g. seven weeks after the patient has started treatment), 3 month follow-up
  Given that this is an intervention study we are assessing changes in outcome over time.

CONTACTS AND LOCATIONS:
Overall Officials: Vendela Zetterqvist, Ph D, Principal Investigator — Uppsala University Hospital
Locations (1):
- Uppsala University Hospital, Uppsala, Uppsala County, Sweden